CLINICAL TRIAL: NCT04206189
Title: Effect of Preoperative Oral Carbohydrates on the Insulin Resistance of Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2019-1014
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Old Age

STUDY DESIGN:
Intervention Model Description: Randomly selected patients of the carbohydrate group are given oral carbohydrate (400ml) 2-3 hours before surgery. In contrast, patients in the control group are fasted water 2 hours before surgery.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate group (Active Comparator)
  Interventions: Dietary Supplement: carbohydrate group - carbohydrate (400ml)
- Control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: carbohydrate group - carbohydrate (400ml) — Randomly selected patients of the carbohydrate group are given oral carbohydrate (400ml) 2-3 hours before surgery. In contrast, patients in the control group are fasted water 2 hours before surgery according to the standard protocol.
  Arms: Carbohydrate group

SUMMARY:
Postoperative cognitive dysfunction (POCD) is more common in older patients, and increased insulin resistance is an important factor for POCD. Fasting before surgery is performed to reduce the incidence of pulmonary aspiration after anesthesia. However, prolonged fasting increases insulin resistance. Recently, it is recommended to minimize fasting times and consume carbohydrate drinks before surgery. Therefore, the investigators investigate whether preoperative carbohydrate drinks can reduce insulin resistance in the elderly patients. Fifty patients (age>65 years) scheduled for arthroplasty will be divided into carbohydrate (n=28) and control (n=28) groups. Randomly selected patients of the carbohydrate group are given 400ml of 12.8 g/100 ml carbohydrate beverage 2-3 hours before their scheduled operation. In contrast, patients in the control group are fasted from water 2 h before surgery according to standard protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing arthroplasty
2. age>65 years

Exclusion Criteria:

1. The subject is a foreigner or illiterate
2. Patients with gastroesophageal reflux disease, gastric emptying disorders, inflammatory bowel disease, or previous treatment for intra-abdominal cancer
3. Patients with chronic renal disease or severe cardiovascular disease
4. HbA1c >69 mmol/mol or BMI >30 kg/m2
5. A duration of ≥5 h between consumption of CHO and initiation of surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Before anesthesia
  Insulin resistance index = glucose x insulin/22.5
Insulin resistance | 1 hour after surgery
  Insulin resistance index = glucose x insulin/22.5

SECONDARY OUTCOMES:
glycemic variability | Before anesthesia
  Coefficient of glucose variability =SD/mean x 100 (%)
glycemic variability | 5 minutes after anesthesia
  Coefficient of glucose variability =SD/mean x 100 (%)
glycemic variability | 1 hour after surgery
  Coefficient of glucose variability =SD/mean x 100 (%)
glycemic variability | 10 minutes after admission of recovery room
  Coefficient of glucose variability =SD/mean x 100 (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine , Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He X, Long G, Quan C, Zhang B, Chen J, Ouyang W. Insulin Resistance Predicts Postoperative Cognitive Dysfunction in Elderly Gastrointestinal Patients. Front Aging Neurosci. 2019 Aug 8;11:197. doi: 10.3389/fnagi.2019.00197. eCollection 2019. PMID 31440156
- [Background] Tang N, Jiang R, Wang X, Wen J, Liu L, Wu J, Zhang C. Insulin resistance plays a potential role in postoperative cognitive dysfunction in patients following cardiac valve surgery. Brain Res. 2017 Feb 15;1657:377-382. doi: 10.1016/j.brainres.2016.12.027. Epub 2016 Dec 31. PMID 28048971
- [Derived] Choi YS, Cho BW, Kim HJ, Lee YS, Park KK, Lee B. Effect of Preoperative Oral Carbohydrates on Insulin Resistance in Older Adults Who Underwent Total Hip or Knee Arthroplasty: A Prospective Randomized Trial. J Am Acad Orthop Surg. 2022 Oct 15;30(20):971-978. doi: 10.5435/JAAOS-D-21-00656. Epub 2022 May 13. PMID 35576534